CLINICAL TRIAL: NCT06557525
Title: Focused Research On Neurofeedback Therapy In Eradicating Depression (FRONTIER)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNB Sumiyoshi Jinja Mae Clinic (Other)
Collaborators: Universal Brain, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: frontier
Record Dates: First submitted 2024-07-21; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurofeedback (Experimental)
  Interventions: Behavioral: Neurofeedback

INTERVENTIONS:
Behavioral: Neurofeedback — Subjects will receive neurofeedback training by visual stimulation using a software program on a PC or tablet (monitor) with reference to EEG data acquired with a portable electroencephalograph (EEG) to provide feedback on the state of the DLPFC in the brain. The DLPFC status of the subject's brain is then fed back to the subject to continue stimulating the subject's reward system. Before and after these neurofeedback training sessions, fMRI imaging will be performed to confirm changes in brain activity.

SUMMARY:
This is an exploratory study to test the efficacy of a novel EEG neurofeedback method in depressed patients. The investigators will measure the change in depressive symptoms before and after the intervention of the novel EEG neurofeedback method using the Depression Rating Scale (primary endpoint). In addition, The investigators will measure the changes in brain activity before and after the intervention using fMRI, and compare the changes in depressive symptoms over the treatment period (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults (at least 18 years old at the time consent is obtained)
* 2. Major depressive episode as defined by the diagnostic criteria of the DSM 5
* 3. One of the following

  1. Hamilton Depression Rating Score (HDRS 17) of 19 or higher
  2. Montgomery Asberg Depression Rating Scale score of 20 or higher
  3. Any other patient deemed appropriate by the PI (subprincipal investigator)
* 4. With respect to taking antidepressants, any of the following

  1. not taking antidepressants
  2. If taking antidepressants, willingness to continue them for the duration of the program.
* 5. If receiving psychotherapy, agree to continue the same psychotherapy for the duration of study participation
* 6. Have treated by a psychiatrist
* 7. Written informed consent
* 8. No planned change in employment status after the study begins

Exclusion Criteria:

* 1. High risk of suicide, such as suicidal ideation or suicide attempts
* 2. History of hospitalization for depression or suicidal behavior
* 3. Comorbid addictions (drugs, alcohol) or history of addictions
* 4. Organic brain disease (e.g., moderate or severe intracranial organic lesions or neurodegenerative disease)
* 5. History of seizures or epilepsy
* 6. Has a serious or unstable physical disease
* 7. Difficulty or inappropriateness/contraindication to MRI imaging
* 8. Pregnant women or unwilling to practice contraception during the study
* 9. Participating in another clinical trial at the same time, or have participated in a clinical trial within the past 90 days, or are scheduled to participate in another clinical trial during the study period, and the principal (sub)investigator determines that participation in another clinical trial may interfere with the results of this study
* 10. Other cases in which the principal investigator (or subinvestigator) determines that it is difficult to conduct this study safely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
HAMD21 change after intervention | 4 weeks after the start of the intervention
  HAMD21(Hamilton Depression Rating Scale, 21-item version) score change compared to baseline.

SECONDARY OUTCOMES:
HAMD21 compared to baseline | 2 and 4 weeks after the start of the intervention and 4, 12, and 24 weeks after the end of the intervention
  HAMD21(Hamilton Depression Rating Scale, 21-item version) score compared to baseline.
MADRS compared to baseline | 2 and 4 weeks after the start of the intervention and 4, 12, and 24 weeks after the end of the intervention
  MADRS(Montgomery Åsberg Depression Rating Scale) score compared to baseline.
SDS compared to baseline | 2 and 4 weeks after the start of the intervention and 4, 12, and 24 weeks after the end of the intervention
  SDS(Self-rating Depression Scale) score compared to baseline.
HAMD21 after intervention | 4 weeks after the start of the intervention
  HAMD21(Hamilton Depression Rating Scale, 21-item version) score
MADRS after intervention | 4 weeks after the start of the intervention
  MADRS(Montgomery Åsberg Depression Rating Scale) score
HAMD21 response rate | 8 weeks after the start of the intervention
  HAMD21(Hamilton Depression Rating Scale, 21-item version) response rate (>=50% reduction)
HAMD21 remission rate | 8 weeks after the start of the intervention
  HAMD21(Hamilton Depression Rating Scale, 21-item version) remission rate (<=7 points)
duration of remission after the end of the intervention | up to 24 weeks after the end of the intervention
  duration of remission if remission occurred after the end of the intervention in HAMD21(Hamilton Depression Rating Scale, 21-item version)
Quality of life assessment (EQ-5D-3L) | 2 and 4 weeks after the start of the intervention and at 4, 12 and 24 weeks after the end of the intervention
  Quality of life assessment (EQ-5D-3L(EuroQol 5 dimensions 3-level))
PHQ-9 score | 2 and 4 weeks after the start of the intervention and at 4, 12, and 24 weeks after the end of the intervention
  PHQ-9(Patient Health Questionnaire-9) score
changes in brain activity | 2 and 4 weeks after the start of the intervention
  EEG data acquired with a portable electroencephalograph (EEG) to provide feedback on the state of the DLPFC in the brain

CONTACTS AND LOCATIONS:
Locations (1):
- UNB Sumiyoshi Jinja Mae Clinic, Fukuoka, Japan